CLINICAL TRIAL: NCT03517852
Title: Intravital Microscopy (IVM) in Patients With Peritoneal Carcinomatosis (PC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emmanuel M. Gabriel, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-009823
Record Dates: First submitted 2018-04-13; First posted 2018-05-08 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Masking Description: This is an open-label, non-randomized, single center, study of IVM observation in conjunction with fluorescein and ICG in subjects with peritoneal carcinomatosis undergoing CRS-HIPEC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Determine the feasibility and clinical utility of performing Human Intravital Microscopy (HIVM) in patients with peritoneal carcinomatosis during standard course of treatment (cytoreductive surgery with hyperthermic intraperitoneal chemotherapy, or CRS-HIPEC).
  Interventions: Device: Human Intravital Microscopy

INTERVENTIONS:
Device: Human Intravital Microscopy — Intravital microscopy (IVM) allows real-time, direct visualization of microscopic blood vessels and calculation of blood flow.

SUMMARY:
This study will investigate the tumor-associated vasculature of patients with peritoneal carcinomatosis, or cancer that spreads along the inner abdominal lining. The investigators will use a technology known as intravital microscopy (IVM) in order to visualize in real-time the tumor-associated vessels of peritoneal disease. The IVM observations may determine if an individual patient's tumor vessels would be amenable to receiving systemic therapy, based on the functionality of the vessels.

DETAILED DESCRIPTION:
Primary objective(s): To determine the feasibility and clinical utility of performing HIVM in patients with peritoneal carcinomatosis during standard course of treatment (cytoreductive surgery with hyperthermic intraperitoneal chemotherapy, or CRS-HIPEC).

Secondary objective(s):

1. Compare the microscopic observation of the tumor-associated vessels with normal tissue (peritoneal surface) in each individual subject.
2. Correlate the microscopic observations of the tumor-associated vessels with pathologic grade of tumor implants.
3. Correlate the microscopic observation of the microvasculature with tumor-specific and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Have an ECOG Performance Status of ≤ 2. Refer to Appendix C.
3. Have measurable disease in the peritoneum by direct visualization (visible lesion typically > 0.5 cm in maximal diameter).
4. Carcinomatosis that meets indications for CRS-HIPEC.
5. Subject must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
6. A negative skin-prick test to fluorescein.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations.
2. Renal dysfunction as defined as a GFR < 45.
3. Liver dysfunction as defined by Child-Pugh score > 5, or LFT's 1.5x above normal range.
4. Any known allergy or prior reaction to fluorescein or ICG or a positive skin prick test to fluorescein.
5. Pregnant or nursing female subjects, determined preoperatively with a urine pregnancy test.
6. Unwilling or unable to follow protocol requirements.
7. Any condition which in the Investigators' opinion deems the patient unsuitable (e.g., abnormal EKG).
8. Any condition that excludes CRS-HIPEC as the standard of care for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Tumor vessel identification (# tumor vessels visualized per high power field) | 15-20 minutes
  Identify and measure vessels associated with peritoneal tumor implants
Tumor vessel density (# tumor vessels per square cm area observed) | 15-20 minutes
  Determine vessel density per 10x field
Fluorescent dye uptake (# tumor vessels with fluorescent dye uptake and # tumor vessels without dye uptake) | 15-20 minutes
  Visualize vital dyes within the vessels [fluorescein and indocyanine green (ICG)]
Tumor blood flow (velocity, mm/sec) | 15-20 minutes
  Calculate the blood flow velocity of the vessels and tissue penetration of fluorescent dyes as markers of vessel permeability.

SECONDARY OUTCOMES:
Post-operative comparison of the microvasculature of peritoneal carcinomatosis with normal tissue (peritoneum) | 15-20 minutes
  The investigators will compare the microvasculature of peritoneal carcinomatosis with normal tissue (peritoneum) in each individual subject using vessel characteristics (diameters, vessel density, detection of intravital dye and flow rates).
Post-operative correlation of the microvasculature with pathologic features of the tumor implants (i.e. tumor grade) at the time of the final pathology report (5-7 days after surgery). | 5-7 days
  The investigators will determine if there is a correlation between the microvasculature with pathologic features of the tumor implants (i.e. tumor grade) at the time of the final pathology report (5-7 days after surgery).
Post-operative correlation of the microscopic observation of the tumor microvasculature tumor-specific and overall survival. | 5 years
  The investigators will determine if there is a correlation between the microscopic observation of the tumor microvasculature tumor-specific and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel M Gabriel, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher DT, Chen Q, Skitzki JJ, Muhitch JB, Zhou L, Appenheimer MM, Vardam TD, Weis EL, Passanese J, Wang WC, Gollnick SO, Dewhirst MW, Rose-John S, Repasky EA, Baumann H, Evans SS. IL-6 trans-signaling licenses mouse and human tumor microvascular gateways for trafficking of cytotoxic T cells. J Clin Invest. 2011 Oct;121(10):3846-59. doi: 10.1172/JCI44952. Epub 2011 Sep 19. PMID 21926464
- [Background] Fisher DT, Muhitch JB, Kim M, Doyen KC, Bogner PN, Evans SS, Skitzki JJ. Intraoperative intravital microscopy permits the study of human tumour vessels. Nat Commun. 2016 Feb 17;7:10684. doi: 10.1038/ncomms10684. PMID 26883450
- [Background] Nagy JA, Chang SH, Shih SC, Dvorak AM, Dvorak HF. Heterogeneity of the tumor vasculature. Semin Thromb Hemost. 2010 Apr;36(3):321-31. doi: 10.1055/s-0030-1253454. Epub 2010 May 20. PMID 20490982
- [Background] Nagy JA, Chang SH, Dvorak AM, Dvorak HF. Why are tumour blood vessels abnormal and why is it important to know? Br J Cancer. 2009 Mar 24;100(6):865-9. doi: 10.1038/sj.bjc.6604929. Epub 2009 Feb 24. PMID 19240721
- [Background] Abdollahi A, Folkman J. Evading tumor evasion: current concepts and perspectives of anti-angiogenic cancer therapy. Drug Resist Updat. 2010 Feb-Apr;13(1-2):16-28. doi: 10.1016/j.drup.2009.12.001. Epub 2010 Jan 12. PMID 20061178
- [Background] Fukumura D, Duda DG, Munn LL, Jain RK. Tumor microvasculature and microenvironment: novel insights through intravital imaging in pre-clinical models. Microcirculation. 2010 Apr;17(3):206-25. doi: 10.1111/j.1549-8719.2010.00029.x. PMID 20374484
- [Background] Skitzki JJ, Chen Q, Wang WC, Evans SS. Primary immune surveillance: some like it hot. J Mol Med (Berl). 2007 Dec;85(12):1361-7. doi: 10.1007/s00109-007-0245-7. Epub 2007 Aug 18. PMID 17704903
- [Background] Jain RK, Munn LL, Fukumura D. Dissecting tumour pathophysiology using intravital microscopy. Nat Rev Cancer. 2002 Apr;2(4):266-76. doi: 10.1038/nrc778. PMID 12001988
- [Background] Murooka TT, Mempel TR. Multiphoton intravital microscopy to study lymphocyte motility in lymph nodes. Methods Mol Biol. 2012;757:247-57. doi: 10.1007/978-1-61779-166-6_16. PMID 21909917
- [Background] Entenberg D, Kedrin D, Wyckoff J, Sahai E, Condeelis J, Segall JE. Imaging tumor cell movement in vivo. Curr Protoc Cell Biol. 2013 Mar;Chapter 19:19.7.1-19.7.19. doi: 10.1002/0471143030.cb1907s58. PMID 23456602
- [Background] McLaughlin RA, Scolaro L, Robbins P, Hamza S, Saunders C, Sampson DD. Imaging of human lymph nodes using optical coherence tomography: potential for staging cancer. Cancer Res. 2010 Apr 1;70(7):2579-84. doi: 10.1158/0008-5472.CAN-09-4062. Epub 2010 Mar 16. PMID 20233873
- [Background] Patsialou A, Bravo-Cordero JJ, Wang Y, Entenberg D, Liu H, Clarke M, Condeelis JS. Intravital multiphoton imaging reveals multicellular streaming as a crucial component of in vivo cell migration in human breast tumors. Intravital. 2013 Apr 1;2(2):e25294. doi: 10.4161/intv.25294. PMID 25013744
- [Background] Franko J, Shi Q, Goldman CD, Pockaj BA, Nelson GD, Goldberg RM, Pitot HC, Grothey A, Alberts SR, Sargent DJ. Treatment of colorectal peritoneal carcinomatosis with systemic chemotherapy: a pooled analysis of north central cancer treatment group phase III trials N9741 and N9841. J Clin Oncol. 2012 Jan 20;30(3):263-7. doi: 10.1200/JCO.2011.37.1039. Epub 2011 Dec 12. PMID 22162570
- [Background] Glehen O, Gilly FN, Boutitie F, Bereder JM, Quenet F, Sideris L, Mansvelt B, Lorimier G, Msika S, Elias D; French Surgical Association. Toward curative treatment of peritoneal carcinomatosis from nonovarian origin by cytoreductive surgery combined with perioperative intraperitoneal chemotherapy: a multi-institutional study of 1,290 patients. Cancer. 2010 Dec 15;116(24):5608-18. doi: 10.1002/cncr.25356. Epub 2010 Aug 24. PMID 20737573
- [Background] Elias D, Gilly F, Boutitie F, Quenet F, Bereder JM, Mansvelt B, Lorimier G, Dube P, Glehen O. Peritoneal colorectal carcinomatosis treated with surgery and perioperative intraperitoneal chemotherapy: retrospective analysis of 523 patients from a multicentric French study. J Clin Oncol. 2010 Jan 1;28(1):63-8. doi: 10.1200/JCO.2009.23.9285. Epub 2009 Nov 16. PMID 19917863
- [Background] Glehen O, Gilly FN, Arvieux C, Cotte E, Boutitie F, Mansvelt B, Bereder JM, Lorimier G, Quenet F, Elias D; Association Francaise de Chirurgie. Peritoneal carcinomatosis from gastric cancer: a multi-institutional study of 159 patients treated by cytoreductive surgery combined with perioperative intraperitoneal chemotherapy. Ann Surg Oncol. 2010 Sep;17(9):2370-7. doi: 10.1245/s10434-010-1039-7. Epub 2010 Mar 25. PMID 20336386
- [Background] Kalogeromitros DC, Makris MP, Aggelides XS, Mellios AI, Giannoula FC, Sideri KA, Rouvas AA, Theodossiadis PG. Allergy skin testing in predicting adverse reactions to fluorescein: a prospective clinical study. Acta Ophthalmol. 2011 Aug;89(5):480-3. doi: 10.1111/j.1755-3768.2009.01722.x. Epub 2009 Nov 10. PMID 19906081
- [Background] Jaffer FA. Intravital fluorescence microscopic molecular imaging of atherosclerosis. Methods Mol Biol. 2011;680:131-40. doi: 10.1007/978-1-60761-901-7_9. PMID 21153378
- [Background] Munn LL, Padera TP. Imaging the lymphatic system. Microvasc Res. 2014 Nov;96:55-63. doi: 10.1016/j.mvr.2014.06.006. Epub 2014 Jun 21. PMID 24956510
- [Background] Wolfe DR. Fluorescein angiography basic science and engineering. Ophthalmology. 1986 Dec;93(12):1617-20. doi: 10.1016/s0161-6420(86)33521-8. PMID 3808620
- [Background] Bloom JN, Herman DC, Elin RJ, Sliva CA, Ruddel ME, Nussenblatt RB, Palestine AG. Intravenous fluorescein interference with clinical laboratory tests. Am J Ophthalmol. 1989 Oct 15;108(4):375-9. doi: 10.1016/s0002-9394(14)73304-5. PMID 2801858
- [Derived] Gabriel EM, Sukniam K, Popp K, Bagaria SP. Human intravital microscopy in the study of sarcomas: an early trial of feasibility. Front Oncol. 2023 Apr 12;13:1151255. doi: 10.3389/fonc.2023.1151255. eCollection 2023. PMID 37124504
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT03517852/Prot_SAP_001.pdf
  • Informed Consent Form (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03517852/ICF_000.pdf